CLINICAL TRIAL: NCT03172897
Title: Low-dose Dexmedetomidine for Delirium Prevention in Mechanically Ventilated Patients in Intensive Care Unit: a Multicenter, Randomised, Double-blinded, Placebo-controlled Trial
Brief Title: Low-dose Dexmedetomidine in Mechanically Ventilated ICU Patients
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was stopped because of difficulty in recruiting patients (another trial had similar inclusion/exclusion criteria). No patients was recruited in this trial.
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017[1319]
Record Dates: First submitted 2017-04-17; First posted 2017-06-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Adult Disease; Intensive Care Unit Syndrome; Mechanical Ventilation Complication; Delirium; Dexmedetomidine
Keywords: Adult; Intensive care unit; Mechanical ventilation; Delirium; Dexmedetomidine
MeSH Terms: conditions — Disease; Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is infused at a rate of 0.1 ug/kg/h for a maximum of 3 days.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Placebo (normal saline) is infused at a same rate as in the dexmedetomidine group for a maximum of 3 days.
  Interventions: Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is administered as a continuous intravenous infusion at a rate of 0.025 mL/kg per h (0.1 μg/kg per h) from study recruitment in the ICU for no more than 72 hours.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo (normal saline) — Placebo (normal saline) is administered as a continuous intravenous infusion at a rate of 0.025 mL/kg per h from study recruitment in the ICU for no more than 72 hours.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
For patients undergoing mechanical ventilation, light sedation is better than deep sedation for the outcomes, which is manifested as shortened length of ICU stay, shortened duration of mechanical ventilation, and decreased mortality. In a recent study of the investigators, low-dose dexmedetomidine without sedative effects (0.1 ug/kg/h) improved sleep quality and reduced the incidence of delirium in elderly patients admitted to the ICU after surgery. The investigators hypothesize that, for ICU patients with prolonged mechanical ventilation, low-dose dexmedetomidine infusion (0.1 ug/kg/h) may also be effective in decreasing delirium. The purpose of this study is to investigate whether low-dose dexmedetomidine infusion can reduce the incidence of delirium in ICU patients with prolonged duration of mechanical ventilation (>= 24 hours).

DETAILED DESCRIPTION:
Delirium is an acutely occurred and transient brain dysfunction characterized with cognitive dysfunction, lowered consciousness, disturbed attention, abnormal psychoactivity, and disordered sleep-wake rhythm. Delirium is frequent in mechanically ventilated patients in the intensive care unit (ICU), with reported incidences up to 70% or 87%. Possible reasons leading to delirium include the intervention-heavy environment of the ICU, mechanical ventilation and sleep disturbances. The occurrence of delirium is associated with worse outcomes including prolonged mechanical ventilation and ICU stay, increased complications, prolonged hospital stay, higher mortality, and elevated medical expenses. It is also associated with worse long-term outcomes including declined cognitive function, lowered life quality, and elevated long-term mortality.

Dexmedetomidine is a high selective alpha-2 adrenoceptor agonist with anxiolytic, sedative and analgesic effects. When used for sedation in mechanically ventilated patients (dose range 0.2-1.4 ug/kg/h), it reduces the consumption of other sedatives and analgesics, ameliorates the rhythm and structure of sleep, and decreases the occurrence of delirium. In recent studies of the investigators, low-dose dexmedetomidine infusion (0.1 ug/kg/h) ameliorated sleep quality; for elderly patients admitted to the ICU after surgery, prophylactic low-dose dexmedetomidine infusion reduced the incidence of delirium (for patients with mechanical ventilation: 28.8% with placebo vs. 11.5% with dexmedetomidine, P<0.0001; for patients without mechanical ventilation: 15.1% with placebo vs. 6.3% with dexmedetomidine, P=0.014).

For patients undergoing mechanical ventilation, light sedation is better than deep sedation for the outcomes, which is manifested as shortened length of ICU stay, shortened duration of mechanical ventilation, and decreased mortality. Some authors even reported that no sedation (analgesia only) provides better outcome than light sedation, because it further shortens the durations of mechanical ventilation and ICU stay. In the above studies of the investigators, the recruited patients were less severe because the Acute Physiology and Chronic Health Evaluation II (APACHE II) score was low (mean score from 10.2 to 10.6) and the duration of mechanical ventilation was short (median 6.9 hours in the control group). The investigators hypothesize that, for ICU patients with prolonged mechanical ventilation, low-dose dexmedetomidine infusion (0.1 ug/kg/h) may also be effective in improving sleep and decreasing delirium. The purpose of this study is to investigate whether low-dose dexmedetomidine infusion can reduce the incidence of delirium in ICU patients with prolonged duration of mechanical ventilation (>= 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older;
* admitted to the ICU;
* with expected duration of mechanical ventilation of more than 24 hours.

Exclusion Criteria:

* refused to participate;
* aged less than 18 years;
* pregnant;
* preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
* inability to communicate in the preoperative period (coma, profound dementia, or language barrier);
* brain injury or neurosurgery;
* known preoperative left ventricular ejection fraction less than 30%, sick sinus syndrome, severe sinus bradycardia (<50 beats per min [bpm]), or second degree or greater atrioventricular block without pacemaker;
* severe hepatic dysfunction (Child-Pugh class C);
* severe renal dysfunction (undergoing dialysis before surgery);
* less likely to survive for more than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within the first 7 days after enrollment | From enrollment until 7 days.
  Assessment twice daily (in the morning from 0600 h to 1000 h and in the evening from 1800 h to 2000 h) with the Confusion Assessment Method for the ICU (CAM-ICU).

SECONDARY OUTCOMES:
Duration of mechanical ventilation | From enrollment until extubation or 30 days.
  Duration of mechanical ventilation after study enrollment.
Length of stay in the ICU | From enrollment until ICU discharge or 30 days.
  Length of stay in the ICU after study enrollment.
Length of stay in the hospital | From enrollment until hospital discharge or 30 days.
  Length of stay in the hospital after study enrollment.
Occurrence of non-delirium complications | From enrollment until 30 days.
  Occurrence of complications other than delirium after study enrollment.
All-cause 30-day mortality | On the 30th day after enrollment.
  All-cause 30-day mortality after study enrollment.
30-day cognitive function | On the 30th day after enrollment.
  Assessed with the Telephone Interview of Cognitive Status-Modified (TICS-m).
30-day life quality | On the 30th day after enrollment.
  Assessed with the WHOQOL-Bref.

OTHER OUTCOMES:
Pain intensity | From enrollment until 7 days.
  Assessed twice daily (in the morning from 0600 h to 1000 h and in the evening from 1800 h to 2000 h) with the Numeric Rating Scale (NRS, an 11 point scale where 0 indicated no pain and 10 indicated the worst possible pain).
Subjective sleep quality | From enrollment until 7 days.
  Assessed in the morning with the NRS (an 11 point scale where 0 indicated the best possible sleep and 10 indicated the worst possible sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nedergaard HK, Jensen HI, Stylsvig M, Lauridsen JT, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients recieving mechanical ventilation - effects on long-term cognitive function: Study protocol for a randomized controlled trial, a substudy of the NONSEDA trial. Trials. 2016 Jun 1;17(1):269. doi: 10.1186/s13063-016-1390-5. PMID 27250658
- [Background] Nedergaard HK, Jensen HI, Lauridsen JT, Sjogaard G, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation--effects on physical function: study protocol for a randomized controlled trial: a substudy of the NONSEDA trial. Trials. 2015 Jul 23;16:310. doi: 10.1186/s13063-015-0856-1. PMID 26201718
- [Background] Toft P, Olsen HT, Jorgensen HK, Strom T, Nibro HL, Oxlund J, Wian KA, Ytrebo LM, Kroken BA, Chew M. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation (NONSEDA Trial): study protocol for a randomised controlled trial. Trials. 2014 Dec 20;15:499. doi: 10.1186/1745-6215-15-499. PMID 25528350
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Background] Porhomayon J, Joude P, Adlparvar G, El-Solh AA, Nader ND. The Impact of High Versus Low Sedation Dosing Strategy on Cognitive Dysfunction in Survivors of Intensive Care Units: A Systematic Review and Meta-Analysis. J Cardiovasc Thorac Res. 2015;7(2):43-8. doi: 10.15171/jcvtr.2015.10. PMID 26191390
- [Background] Balzer F, Weiss B, Kumpf O, Treskatsch S, Spies C, Wernecke KD, Krannich A, Kastrup M. Early deep sedation is associated with decreased in-hospital and two-year follow-up survival. Crit Care. 2015 Apr 28;19(1):197. doi: 10.1186/s13054-015-0929-2. PMID 25928417
- [Background] Treggiari MM, Romand JA, Yanez ND, Deem SA, Goldberg J, Hudson L, Heidegger CP, Weiss NS. Randomized trial of light versus deep sedation on mental health after critical illness. Crit Care Med. 2009 Sep;37(9):2527-34. doi: 10.1097/CCM.0b013e3181a5689f. PMID 19602975
- [Background] Hughes CG, Girard TD, Pandharipande PP. Daily sedation interruption versus targeted light sedation strategies in ICU patients. Crit Care Med. 2013 Sep;41(9 Suppl 1):S39-45. doi: 10.1097/CCM.0b013e3182a168c5. PMID 23989094
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Xia ZQ, Chen SQ, Yao X, Xie CB, Wen SH, Liu KX. Clinical benefits of dexmedetomidine versus propofol in adult intensive care unit patients: a meta-analysis of randomized clinical trials. J Surg Res. 2013 Dec;185(2):833-43. doi: 10.1016/j.jss.2013.06.062. Epub 2013 Jul 24. PMID 23910886
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Wunsch H, Kahn JM, Kramer AA, Wagener G, Li G, Sladen RN, Rubenfeld GD. Dexmedetomidine in the care of critically ill patients from 2001 to 2007: an observational cohort study. Anesthesiology. 2010 Aug;113(2):386-94. doi: 10.1097/ALN.0b013e3181e74116. PMID 20613466
- [Background] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955
- [Background] Djaiani G, Silverton N, Fedorko L, Carroll J, Styra R, Rao V, Katznelson R. Dexmedetomidine versus Propofol Sedation Reduces Delirium after Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2016 Feb;124(2):362-8. doi: 10.1097/ALN.0000000000000951. PMID 26575144
- [Background] Mo Y, Zimmermann AE. Role of dexmedetomidine for the prevention and treatment of delirium in intensive care unit patients. Ann Pharmacother. 2013 Jun;47(6):869-76. doi: 10.1345/aph.1AR708. PMID 23719785
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Scott BK. Disruption of Circadian Rhythms and Sleep in Critical Illness and its Impact on the Development of Delirium. Curr Pharm Des. 2015;21(24):3443-52. doi: 10.2174/1381612821666150706110656. PMID 26144937
- [Background] Francis J, Kapoor WN. Prognosis after hospital discharge of older medical patients with delirium. J Am Geriatr Soc. 1992 Jun;40(6):601-6. doi: 10.1111/j.1532-5415.1992.tb02111.x. PMID 1587979